CLINICAL TRIAL: NCT04043468
Title: Effects of an Action Support Component in Audit and Feedback Interventions With Primary Care Nursing Teams: A Pragmatic Trial
Brief Title: Audit and Feedback Interventions With Primary Care Nursing Teams
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: CR-CSSS Champlain-Charles-Le Moyne (Other)
Responsible Party: Principal Investigator, Emilie Dufour, Principal Investigator, CR-CSSS Champlain-Charles-Le Moyne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CharlesLeMoyne
Record Dates: First submitted 2019-07-20; First posted 2019-08-02 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Nurse's Role
Keywords: audit and feedback; process indicators; quality

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Improved A&F intervention (Experimental): Two feedback sessions and four structured focus groups
  Interventions: Other: Audit and feedback
- Standard A&F intervention (Active Comparator): Two feedback sessions
  Interventions: Other: Audit and feedback

INTERVENTIONS:
Other: Audit and feedback — Audit and feedback (A&F) is an intervention that aims to improve professionals practices by providing professionals with a summary of their performance over a period of time.

SUMMARY:
Audit and feedback (A&F) aims to improve practices by providing professionals with a summary of their performance. A major limitation to its effectiveness is a persistent intention-action gap following the feedback that prevents the translation of planned actions into concrete changes in practice. In nursing, the lack of coordination within nursing teams contributes to this gap and therefore limits their capacity for action. The objective of this study is to evaluate the effects of an A&F intervention enhanced with an action support component on the primary care nursing teams' capacity to improve performance compared to a standard A&F intervention.

A pragmatic cluster randomised controlled trial with analysis of implementation fidelity will be conducted. Four nursing organizations will receive standard A&F, while the other four will receive A&F with a support component. We will measure performance using clinical administrative data from an electronic database based on wound care episodes. Performance indicators will be measured 3 times: at the beginning of the study (T1), after 6 months (T2) and after 12 months (T3). The feedback meetings will take place between times 1 and 2, then between times 2 and 3. The intervention group will receive the support component in the form of structured focus groups in addition to the feedback meetings. Changes in rates of seven nursing-sensitive indicators (continuity, planning and adjusting of the treatment plan, initial assessment, education, frequency and number of consultations and duration of episodes) will be measured to evaluate the effects of A&F on performance.

The results are expected to inform of the effectiveness of A&F in order to improve its design and deployment. The potential impact on the improvement of practices is significant, considering that wound care is one of the main conditions in primary care for which nursing staff have a high degree of autonomy.

DETAILED DESCRIPTION:
Audit and feedback (A&F) is an intervention that aims to improve professionals practices by providing professionals with a summary of their performance over a period of time. A&F has 1) an audit phase, in which performance indicators are measured and 2) a feedback phase, in which the indicators are reported to the professionals to encourage reflexive practice and determine an action plan. Although its effectiveness has been demonstrated, it is widely accepted that this type of intervention is highly variable and that its design has considerable room for improvement. A major limitation to the effectiveness of A&F is a persistent intention-action gap encounters by professionals following the feedback. This gap prevents the translation of planned actions into concrete changes in practice. In nursing, an aspect that contributes to this gap is a lack of coordination of actions within nursing teams, which limits their capacity for collective action.

Purpose and objectives: The purpose of this study is to evaluate the effects of an A&F intervention enhanced with an action support component on the primary care nursing teams' capacity to improve performance compared to a standard A&F intervention. This study has two specific objectives: 1) to measure the effects of the addition of structured focus groups during an enhanced A&F intervention on the performance levels of the process and outcome indicators compared with the measured effects of standard A&F intervention; and 2) to analyze the effects of the implementation fidelity of the standard and enhanced A&F interventions on the effectiveness of A&F.

Method: A pragmatic cluster randomised controlled trial with analysis of implementation fidelity will be conducted. Eight primary care nursing organizations will be included. Four of them will receive a standard A&F intervention, while the remaining four will receive an AF intervention with a support component. Performance will be measured using clinical administrative data from an electronic database currently used to compile statistics on the services provided and the users of Local community service centers (CLSC) in Quebec. Performance will be measured from wound care episodes of patients who had a follow-up during the study period. Four process indicators (continuity, planning and adjusting of the treatment plan, initial assessment and education) and three outcome indicators (frequency and number of consultations and duration of episodes) sensitive to nursing care will be measured 3 times: at the beginning of the study (T1), after 6 months (T2) and after 12 months (T3). The feedback meetings will take place between times 1 and 2, then between times 2 and 3. The intervention group will receive the support component in the form of structured focus groups in addition to the feedback meetings, twice between each of the time periods. Models of generalized estimating equations will be adjusted to analyze differences in performance in each group. An analysis of implementation fidelity will be conducted in parallel of the pragmatic trial using grids of observations in each of the settings

ELIGIBILITY:
Inclusion Criteria:

* The inclusion and exclusion criteria are at two levels: 1) primary care organizations and 2) wound care episodes that will be used to measure performance improvement. Nursing organizations that offer services seven days a week will be included so that they can measure all the selected indicators and use the I-CLSC software in their daily practice. Wound care episodes with a minimum duration of 7 days and an episode start during the measurement period will be included. These two criteria are applied in order to measure the seven indicators.

Exclusion Criteria:

* Wound care episodes in palliative care will be excluded, as the indicators were selected for episodes of wound care with healing potential. Such episodes are identifiable by codes in the database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-02 (Estimated); Primary Completion 2023-09-02 (Estimated); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
Continuity | Change from baseline continuity at 6 and 12 months.
  Percentage of care episodes in which at least 50 % of the consultations are provided by the same professional
Planning and adjusting of the treatment plan | Change from baseline Planning and adjusting of the treatment plan at 6 and 12 months.
  Percentage of care episodes in which at least 75 % of the consultations are with an RN
Education | Change from baseline Education at 6 and 12 months.
  Percentage of care episodes in which at least one education session is provided
Initial assessment | Change from baseline Initial assessment at 6 and 12 months.
  Percentage of care episodes in which a RN performs a wound assessment in the first consultation
Frequency | Change from baseline Frequency at 6 and 12 months.
  Percentage of care episodes with no more than three consultations per week as of the second week
Duration | Change from baseline Duration at 6 and 12 months.
  Percentage of care episodes lasting 42 days or less
Intensity | Change from baseline Intensity at 6 and 12 months.
  Percentage of care episodes with no more than 22 consultations

IPD SHARING:
Plan to Share IPD: No